CLINICAL TRIAL: NCT04331119
Title: Phase II Trial With Safety Lead in of Duvelisib Maintenance After Autologous Stem Cell Transplant in T-Cell Lymphomas
Brief Title: Duvelisib Maintenance After Autologous Stem Cell Transplant in T-Cell Lymphomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202005165
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Duvelisib Maintenance (Experimental): * Duvelisib maintenance at 25 mg PO BID after count recovery (approximately 30 days after transplant) for one year. If the patient is in a complete remission at day +100, with no evidence of disease on PET/CT, then the dosing schedule of duvelisib may be changed to 25 mg BID for 14 days, then 14 days off in 28 day cycles (at the treating physician's discretion). If the patient has residual disease, duvelisib will continue at 25 mg BID until they have a negative PET CT. PET CTs will be completed every 3 months for patients with residual disease. Duvelisib maintenance will be continued for one year post-transplant.
  * Starting on 06/10/2021, all new participants will be enrolled to take 25 mg BID of duvelisib on days 1-14 of a 28 day cycle.
  Interventions: Drug: Duvelisib; Procedure: Peripheral blood draw

INTERVENTIONS:
Drug: Duvelisib — SecuraBio will supply duvelisib
  Other Names: Copiktra
Procedure: Peripheral blood draw — -Prior to transplant, cycle 1 day 1 of duvelisib, and at the time of all imaging studies

SUMMARY:
The investigators hypothesize that duvelisib maintenance after autologous stem cell transplant in patients with T-cell lymphomas will be safe and well tolerated, and will improve progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T cell non-Hodgkin lymphoma, T cell lymphomas included are peripheral T cell lymphoma not otherwise specified, angioimmunoblastic T cell lymphoma, and systemic anaplastic large cell lymphoma.
* Eligible for autologous stem cell transplantation as determined by the treating physician or completed autologous transplant within the last 30 days.
* At least 18 years of age at time of enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ function as defined below:

  * Serum creatinine ≤ 1.5 times institutional upper limit of normal (IULN)
  * Total bilirubin ≤ 1.5 x IULN. Patients with Gilbert's Syndrome may have a bilirubin > 1.5 x IULN
  * Hemoglobin ≥ 8.0 g/dL
  * Absolute neutrophil count ≥ 1.0 x 109/L
  * Platelet count ≥ 75 x 109/L
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
* Women of childbearing potential and men must agree to use highly effective contraception prior to study entry and for the duration of study participation and for 3 months after the last dose of duvelisib. Negative serum β human chorionic gonadotropin (βHCG) pregnancy test within 7 days before first treatment is required if the patient is a woman of childbearing potential.
* Participants or a participant's legally authorized representative must be able to understand and willing to sign an IRB approved written informed consent document

Exclusion Criteria:

* Currently receiving any other experimental therapy or has received experimental therapy within 4 weeks prior to study treatment
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to duvelisib or other agents used in the study.
* Prior history of drug-induced colitis or drug-induced pneumonitis
* History of concurrent interstitial lung disease or severely impaired lung function
* History of chronic liver disease or veno-occlusive disease
* History of tuberculosis within 2 years prior to enrollment
* Administration of a live or live attenuated vaccine within 6 weeks of first duvelisib dose
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine) or systemic steroids > 20 mg of prednisone (or equivalent) per day
* Ongoing treatment for systemic bacterial, fungal, or viral infections at screening.

Note: patients on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded is all other inclusion/exclusion criteria are met

* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV) at screening
* Infection with HBV, HCV. Subjects with a positive HBsAg or HCV Ab on pre-transplant infection screening will be excluded. Subjects with a positive HBcAb must have negative HBV DNA to be eligible and must be periodically monitored for HBV reactivation by institutional guidelines.
* Baseline QTcF > 500 milliseconds. This does not apply to subjects with right or left bundle branch blocks
* Concurrent active malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix, bladder cancer, or prostate cancer not requiring treatment.
* Clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea,vomiting, or any other condition that will interfere significantly with drug absorption
* Concurrent administration of medications or foods that are strong inhibitors or inducers of cytochrome P450 3A (CYP3A). No prior use within 2 weeks before the start of study intervention.
* Active cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection (i.e., subjects with detectable viral load)
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or a pacemaker within the last 6 months prior to screening.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or unstable cardiac arrhythmia.
* Pregnant or breastfeeding.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended. Recommend exclusion of specific ART agents based on predicted drug-drug interactions (i.e. concurrent strong CYP3A4 inhibitors (ritonavir and cobicistat) or inducers (efavirenz) are contraindicated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  The PFS time will be calculated as the duration of time from autologous stem cell transplant (day 0) to the date of earliest progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Safety and tolerabilty as measured by number of study treatment related adverse events | From start of treatment through 30 days after last dose of duvelisib (estimated to be 13 months)
  -Adverse events will be assessed using CTCAE v5.0 criteria
Safety and tolerabilty as measured by discontinuations due to treatment-related adverse events | From start of treatment through 30 days after last dose of duvelisib (estimated to be 13 months)
Overall response rate (ORR) | 100 days after transplant
  -Defined as the percentage of patients with a confirmed complete or partial response, monitored with PET/CT scans.
Overall survival (OS) | 2 years
  -Defined as the duration of time from the date of first dose of study treatment to death from any cause. Patients who are alive by the data cutoff date will be censored at the last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu